# UNIVERSITY OF CALIFORNIA, SAN FRANCISCO ASSENT TO BE IN RESEARCH

**Study Title:** The Technology-based Resources to increase Uptake of Sexual health services for Teens (TRUST) Study

This is a research study, and you do not have to take part. This study is conducted by Dr. Jyu-Lin Chen, Associate Professor at UCSF Department of Family Health Care Nursing and Dr. Kimberly Koester, Assistant Professor at UCSF Department of Medicine. The research assistant will explain this study to you. If you have any questions, you may ask the research assistant.

You are being asked to be in the study because you are a teenager (age 11-17 years old) at one of the clinics, we are working with to develop and test the TRUST intervention.

In this study, the researchers are conducting a study to learn more about how to strengthen the partnerships between adolescents (11-17 year old), their mothers/female guardians and their healthcare providers. The purpose of this study is to seek feedback from teenagers on the TRUST intervention. We want to find out if we can help improve your health by encouraging you to have time alone with your doctor to talk about important topics such as sexual health in private without your parent or guardian in the room.

The Centers of Disease Control is paying for this research. About 40-60 adolescents and their mothers that will take part in this study.

#### What will happen if I take part in this study?

If you agree to be in this study, you will be asked to take part in the following:

- 1. You will attend your well child visit as usual and be asked to take a survey afterwards on spending time alone with your healthcare provider.
- 2. You will be asked to fill out 2 surveys about communication with your parent through the study website (TRUSTSTUDY.UCSF.EDU).
- 3. You will be asked to visit the GritX website at UCSF (https://gritx.org/courses.php)
  - -On the GritX website you will be sent messages with information on spending time alone with your healthcare provider and communicating with your parent.
  - -You will be asked to explore interactive and culturally tailored materials to learn more about sexual health, communication, and spending time alone with your healthcare provider.
- 4. All survey reports will be kept confidential. That means that no one will be told your answers. Not your parents or doctor.

You will contribute about 1-3 hours of time while participating in this study.

# How will my information be used?

Researchers will use your information to conduct this study. Information gathered during this research study will only be used for this study. It will not be shared with other researchers.

# Are there any risks to me or my privacy?

Some of the survey questions may make you feel uncomfortable or raise unpleasant memories. You are free to skip any question.

We will do our best to protect the information we collect from you. Information that identifies you will be kept secure. The survey itself will not include details that directly identify you, such as your name or address. Please do not put this information on your survey. The completed surveys will be kept secure and separate from information that identifies you. Only a small number of researchers will have direct access to completed surveys. If this study is published or presented at scientific meetings, names and other information that might identify you will not be used.

Authorized representatives from the following organizations may review your research data for the purpose of monitoring or managing the conduct of this study:

- Representatives of the University of California
- Representatives of the Centers for Disease Control

#### Are there benefits?

Teenagers participating in this study may learn about sexual health resources and effective communication while taking part in this study.

## Can I say "No"?

Yes, you do not have to take part in the study. If you choose not to be in this study you will not lose any of your regular benefits, and you can still receive medical care from UCSF.

## Are there any payments or costs?

You will not be charged for any of the study's procedures. In return for your time and effort you will receive \$70 gift card after the completion of the study.

## Who can answer my questions about the study?

You can talk with the study researcher about any questions, concerns, or complaints you have about this study. Contact the study researcher(s) Jyu-Lin Chen at 415-502-6015.

If you wish to ask questions about the study or your rights as a research participant to someone other than the researchers or if you wish to voice any problems or concerns you may have about the study, please call the office of the Institutional Review Board at 415-476-1814.

# **CONSENT**

| PARTICIPATION I | N RESEARCH IS VOLUNTARY. |
|---|---|
| You have been given | n copies of this consent form to keep. |
| If you wish to be in this study, please sign below. | |
| Date | Participant's Signature for Consent |
| Date | Person Obtaining Consent |